CLINICAL TRIAL: NCT04010890
Title: Development and Evaluation of Culturally Adapted CBT to Improve Community Mental Health Services for Canadians of South Asian Origin
Brief Title: Development and Evaluation of Culturally Adapted CBT for South Asian Canadians
Acronym: CaCBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Farooq Naeem, Professor, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAddictionMH
Record Dates: First submitted 2019-07-01; First posted 2019-07-08 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Depression; Anxiety
Keywords: culture; cognitive therapy; Canada
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This mixed study will be conducted in 3 phases
  1. Development of culturally adapted CBT for Canadian South Asians through a qualitative study
  2. Testing culturally adapted CBT against standard CBT for efficacy through RCT and economic evaluation
  3. Evaluation of training of therapists in culturally adapted CBT
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally adapted CBT (Experimental): Ca_CBT will be delivered to the experimental group using the newly developed manual . The intervention will be delivered over 8-12 sessions. The Control group will receive standard CBT
  Interventions: Behavioral: Culturally adapted CBT
- Standard CBT (Active Comparator): Participants in this group will receive standard CBT
  Interventions: Behavioral: Culturally adapted CBT

INTERVENTIONS:
Behavioral: Culturally adapted CBT — Culturally adapted CBT for South Asian Canadians
  Other Names: CaCBT

SUMMARY:
As CBT was developed for persons from North America and European background it needs to be adapted for persons from non-Western cultures. This mixed methods study proposes a culturally adapted Cognitive Behavioural Therapy (CA-CBT) model for Canadians of South Asian origin. Beginning with a participatory/qualitative research approach, common themes amongst individuals with depression and/or anxiety, caregivers, healthcare professionals, and community leaders, will divulge basic elements needed to develop a culturally adapted model of cognitive behavioural therapy. The information from the adapted model will be taught to participating therapists who will deliver the therapy in a randomized control trial design, with feasibility testing of the intervention using a quantitative approach. Immediate guidelines will then be developed for use by therapists working with South Asian clients.

DETAILED DESCRIPTION:
Background and Significance:

Canadians of South Asian (SA) origin, defined as individuals with ancestral ties to India, Pakistan, Bangladesh, Sri Lanka, Bhutan, Afghanistan, Maldives and Nepal, comprise the largest racialized group in Canada, amounting to 1.6 million individuals or 5% of the Canadian population and 32% of the Canadian Asian population. This makes them the largest visible minority group in Canada, comprising 25.6% of the visible minority population, followed by East Asian and African-Caribbean Canadians, respectively. The SA Canadians are disproportionately affected by high rates of anxiety and mood disorders, placing those immigrating to Canada at age 17 or younger at a significantly higher risk for this condition compared to immigrants from elsewhere who immigrated at the same age.

The SA Canadians are disproportionately impacted by the social determinants of health, including unemployment, low income, language barriers, low education, low literacy and migration stress. These factors can negatively impact mental health and decrease access to care, thereby increasing mental health inequities. Compared to other ethnocultural groups, SA Canadians with a major depressive episode reported the highest proportion of unmet mental health care needs (48%) and the highest percentage of perceived barriers to the availability of mental health care(33%). Canadians who had a major depressive episode and identified as SA were 85% less likely to seek treatment than Canadians who had experienced the same illness but identified as white. The lower use of mental health services by SA Canadians highlights the inequities in access to appropriate care for these populations.

The Mental Health Commission of Canada (MHCC) recommends improving Canadian mental health care to serve diverse populations with equitable, timely access to appropriate, effective, and evidence-based treatments that attend to unique sociocultural needs (Mental Health Commission of Canada, 2014). The MHCC Case for Diversity report further highlights the necessity for culturally and linguistically relevant services particularly for immigrant, refugee, ethnocultural and racialized populations, such as SA Canadians. In light of the new $5B targeted federal transfer to "improve access to mental health and addiction services and to structured psychotherapy" (Government of Canada, 2016) there is an opportunity to complement efforts to expand the access that adequately address the mental health needs of diverse Canadian populations.

Cognitive Behavioural Therapy in its current form is not suitable for persons from the non-western cultural background. Culturally-adapted Cognitive Behavioural Therapy (Ca_CBT) is an evidence-based practice. CaCBT is more effective than standard CBT and can reduce dropouts from therapy compared with standard CBT. Thus CaCBT can increase access to mental health services and improve outcomes for immigrant, refugee, ethnocultural and racialized populations. Adapting CBT for growing SA populations in Canada will ensure equitable access to effective, culturally-appropriate interventions. Accordingly, this study proposes to develop and evaluate Ca_CBT for depression and anxiety among SA populations in Canada.

Study Objectives:

The primary objective of the study is to develop culturally adapted CBT for South Asian persons with depression and anxiety. Secondary objectives include; (a) testing CaCBT against standard CBT for efficacy and cost-effectiveness, and (b) to test whether training in culturally adapted CBT can improve therapist's cultural competence.

Methods:

This mixed methods study will be conducted in three phases:

Phase 1: Cultural Adaptation of CBT Cultural adaptation of CBT for SA populations in Canada experiencing depression and anxiety using stakeholder consultations and qualitative methodology

Phase 2: Pilot Feasibility Testing of Ca_CBT Pilot test the newly developed Ca_CBT for feasibility, acceptability and effectiveness via quantitative methodology and a randomized controlled trial

Phase 3: Implementation & Evaluation of Ca_CBT Trained therapists working with SA populations to use Ca_CBT with their clients. Evaluate therapist competence in using Ca_CBT as well as client satisfaction with the newly developed therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants, between the ages of 18 - 64
2. who score 8 or more on the Hospital Anxiety and Depression Scale (HADS) Depression Subscale Or on Anxiety Subscale, will be included in the study.

Exclusion Criteria:

1Participants who are dependent on alcohol or drugs (using DSM V criteria) 2. Those with significant cognitive impairment (e.g. intellectual disability or dementia) 3. With active psychosis 4. Participants who have received CBT during the previous 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-07-26 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 36 weeks
  HADS is a 14-item, self-assessment scale designed to measure anxiety and depression. The maximum score is 21 for depression and 21 for anxiety. A score of 8 - 10 suggests the presence of the borderline cases, while a score of 11 - 21 indicates abnormal cases.

SECONDARY OUTCOMES:
WHO DAS 2 (World Health Organization, Disability Assessment Scale, 2nd version) | 36 weeks
  This scale assesses disability due to physical and psychological problems and has been used extensively in various research settings.
Bradford Somatic Inventory | 36 weeks
  The Bradford Somatic Inventory (BSI) enquires about a wide range of somatic symptoms during the previous month and has 45 items. Scores above 21 indicate depression

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Pollock, Study Chair — Center for Addiction and Mental Health
Locations (3):
- Canada (3):
  - Somerset West Mental Health Services, Ottawa
  - Punjabi Health, Toronto
  - Moving Forward, Vancouver

REFERENCES:
- [Derived] Naeem F, Tuck A, Mutta B, Dhillon P, Thandi G, Kassam A, Farah N, Ashraf A, Husain MI, Husain MO, Vasiliadis HM, Sanches M, Munshi T, Abbott M, Watters N, Kidd SA, Ayub M, McKenzie K. Protocol for a multi-phase, mixed methods study to develop and evaluate culturally adapted CBT to improve community mental health services for Canadians of south Asian origin. Trials. 2021 Sep 6;22(1):600. doi: 10.1186/s13063-021-05547-4. PMID 34488853